CLINICAL TRIAL: NCT06588530
Title: Effects of Exposure to Per- and Polyfluoroalkyl Substances (PFAS) on Innate and Adaptive Immune Responses to Tetanus-diphtheria (Td) Vaccination Among Adults in a Community-based Panel Study
Brief Title: PFAS Exposure and Immune Response to Vaccination in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Robert Laumbach MD, MPH, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2024000644
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Innate Inflammatory Response; Vaccination; Diphtheria; Tetanus; Environmental Exposure; Vaccine; Antibodies; Adult; Immunity; Pollution; Exposure
Keywords: PFAS; Perfluoroalkyl substances; Polyfluoroalkyl substances; Vaccine; fluorocarbons; tetanus-diphtheria vaccine; prospective study; Adaptive immunity; innate immunity; PFNA, Perfluorononanoic Acid
MeSH Terms: conditions — Inflammation; Diphtheria; Tetanus | interventions — Diphtheria-Tetanus Vaccine; Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants will be vaccinated during their first study visit using TENIVAC (Tetanus and Diphtheria Toxoids Adsorbed).TENIVAC will be administered intramuscularly as recommended in the subject's deltoid muscle at a dose of 0.5 mL.
  Interventions: Biological: TENIVAC

INTERVENTIONS:
Biological: TENIVAC — TENIVAC (Tetanus and Diphtheria Toxoids Adsorbed) is an active immunization for the prevention of tetanus and diphtheria in persons 7 years of age and older.
  Other Names: Tetanus and Diphtheria Toxoids Adsorbed; Td

SUMMARY:
This clinical trial aims to investigate how exposure to Perfluorononanoic acid (PFNA), a type of per- and polyfluoroalkyl substance (PFAS), affects the immune response to the standard tetanus and diphtheria (Td) vaccine. The study focuses on participants from a community with known prior PFNA exposure through contaminated drinking water. The main question it aims to answer is:

* Does exposure to PFNA weaken the body's initial immune response, leading to lower levels of protective antibodies after vaccination?

Participants will:

* Receive Tetanus and Diphtheria (Td) booster vaccination
* Visit the study office 7 times over a 30-day period
* Have blood and saliva collected at each study visit

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Paulsboro PFAS Health Study
* Provided a blood sample for the Paulsboro PFAS Health Study
* Weigh at least 110 pounds

Exclusion Criteria:

* Currently Pregnant
* History of difficult blood draws
* History of adverse reaction to prior vaccinations
* Currently taking immune suppressants
* Recent dental surgery or dental procedure within 4 weeks of starting study
* Had a Td booster in the past 10 years

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Laumbach, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- EOHSI Paulsboro Office, Paulsboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High PFNA Exposure: Serum Perfluorononanoic acid (PFNA) was previously measured. Participants whose pre-enrollment serum PFNA concentrations were in the higher exposure range, defined as falling within the 4th or 5th quintiles of the PFNA distribution. All participants received a single 0.5 mL intramuscular dose of TENIVAC (Tetanus and Diphtheria Toxoids Adsorbed) at Visit 1. Td-specific IgG concentrations were measured at baseline and 30 days post-vaccination.
- Low PFNA Exposure: Serum Perfluorononanoic acid (PFNA) was previously measured. Participants whose pre-enrollment serum PFNA concentrations were in the lower exposure range, defined as falling within the 1st, 2nd, and 3rd quintiles of the PFNA distribution. All participants received a single 0.5 mL intramuscular dose of TENIVAC (Tetanus and Diphtheria Toxoids Adsorbed) at Visit 1. Td-specific IgG concentrations were measured at baseline and 30 days post-vaccination.
Period: Overall Study
Arm/Group | High PFNA Exposure | Low PFNA Exposure
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High PFNA Exposure | Low PFNA Exposure | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 50.2 [31 to 68] | 49.3 [31 to 70] | 49.75 [31 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 9 | 13
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  Healthy (18.5 - 24.9 *kg/m^2*) | 1 | 2 | 3
  Overweight (25.0 - 29.9 *kg/m^2*) | 4 | 3 | 7
  Obesity (30.0 or above*kg/m^2*) | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Tetanus-diphtheria Specific IgG by PFNA Exposure Category
Description: Quantitative measurement of tetanus and diphtheria specific IgG antibodies in serum collected at baseline (pre-vaccination) and Day 30 post-vaccination. Change is expressed as log₂ transformed fold change: log₂(day30 IgG / baseline IgG). IgG concentrations were measured using commercially available ELISA kits following the manufacturer's instructions. Serum PFNA levels were measured prior to enrollment. IgG was measured at baseline and 30 days post vaccination.
Time Frame: 30 days
Population: All participants with IgG measurements at baseline and Day 30
Measure: Mean (Standard Deviation); unit: log2(fold change)
Arm/Group | High PFNA Exposure | Low PFNA Exposure
Number analyzed (Participants) | 10 | 10
log2(fold change)
  Change in Tetanus IgG | 3.54 (1.83) | 3.39 (1.91)
  Change in Diphtheria IgG | 2.44 (1.47) | 2.43 (1.60)
Statistical Analysis 1: Comparison: High PFNA Exposure vs Low PFNA Exposure; Tetanus; Test type: Other — Log₂ transformed fold change in IgG concentration from baseline to Day 30 was compared between High and Low PFNA exposure groups using the Wilcoxon rank-sum test. A two-tailed significance level of 0.05 was used; p = .85, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.15
Statistical Analysis 2: Comparison: High PFNA Exposure vs Low PFNA Exposure; Diphtheria; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .85, Wilcoxon (Mann-Whitney); Mean Difference (Net) = .01

ADVERSE EVENTS:
Time Frame: 30 days after vaccination
Arm/Group | High PFNA Exposure | Low PFNA Exposure
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT06588530/Prot_SAP_002.pdf
  • Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT06588530/ICF_003.pdf